CLINICAL TRIAL: NCT06084208
Title: A Prospective Investigation to Assess the Diagnostic Yield of Using a Robotic Navigational Bronchoscopy System With Adjunct Real-time Imaging
Brief Title: Assessment of Diagnostic Yield Using a Robotic Navigational Bronchoscopy System With CBCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ISI-ION-EU2-2023
Record Dates: First submitted 2023-09-20; First posted 2023-10-16 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Biopsy; Bronchoscopy
MeSH Terms: conditions — Lung Neoplasms | interventions — Biopsy

STUDY DESIGN:
Intervention Model Description: A prospective, single-center, dual-arm, interventional study, where data from 131 recruited patients undergoing a Robotic Navigational Bronchoscopy System procedure with CBCT are compared to 91 matched Navigation Bronchoscopy with CBCT controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Robotic Navigational Bronchoscopy (Experimental): Patients undergoing biopsy with the Ion Endoluminal System
  Interventions: Device: Biopsy with the Robotic- Ion Endoluminal System with Adjunct Real-time Imaging

INTERVENTIONS:
Device: Biopsy with the Robotic- Ion Endoluminal System with Adjunct Real-time Imaging — Biopsy with the Robotic- Navigational Bronchoscopy System with Cone Beam Computed Tomography (CBCT)

SUMMARY:
The aim of this research study is to evaluate the effectiveness of the ION endoluminal system at reaching and obtaining biopsies from lung nodules when used in combination with 3-dimensional imaging such as CT scans. The learning curve of the procedure will be assessed and data on safety will also be collected.

DETAILED DESCRIPTION:
This is a prospective, interventional, single-centre, dual-arm study which will be conducted in the Netherlands and will involve up to 131 patients undergoing a pulmonary nodule biopsy using the Ion Endoluminal System in conjunction with 3D imaging. Outcomes in these patients will be compared to 91 propensity score matched Cone Beam CT- Navigational Bronchoscopy (CBCT-NB) controls obtained from the site's existing CBCT-NB database.

The objectives of the study are focused on evaluating the procedure learning curve and characteristics of the pulmonary nodule biopsy procedure, including diagnostic yield, rate of tool in nodule, sensitivity for malignancy and safety.

A learning curve analysis will be retrospectively performed to determine when both operators have reached competency with the Ion Endoluminal System. Criteria for passing the learning curve for measuring proficiency in the CUSUM will be diagnostic yield. Additional parameters like tool in lesion and procedure durations will also be monitored.

All subjects will be followed up at 1 week after the procedure. If an adverse event was observed, a 30-day post-procedure visit will also take place. If the biopsy did not provide a diagnosis or did not show cancer and was still under observation, then they will have further follow up at 6 months. Similarly, if the status is unchanged (non-malignant diagnosis) and the nodule is still under observation, a 13 months visit should be completed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is aged 18 years or older at time of consent.
2. Patient is suitable for elective nodule biopsy via bronchoscopy under general anesthesia per Investigator's discretion.
3. Patient has solid or semi-solid pulmonary nodule(s) of ≥6 mm and ≤3 cm in largest dimension (based on pre-procedure CT scan).
4. Pulmonary nodule(s) intended for biopsy during the study procedure is (are) located at least 4 (≥4) airway generations out (trachea = generation 0, e.g. subsegmental bronchi or beyond) based on pre-procedure CT scan.
5. Patient has a moderate to high risk of lung cancer based on clinical, demographic, and radiologic information or with suspected metastatic disease. High risk for malignancy patients are eligible if a biopsy is required or requested prior to intervention.
6. Patient is willing and able to give written informed consent for Clinical Investigation participation.
7. Patient is not legally incapacitated or in a legal/court ordered institution.

Exclusion Criteria:

1. Patient has a lack of fitness or exercise capacity to undergo bronchoscopy under general anesthesia as determined by Investigator prior to procedure.
2. Patient with type 1 pure ground glass opacity target nodule(s) intended for biopsy during study procedure.
3. Presence of bullae(s) with a size of >1 cm on pre-procedure CT scan located in close proximity to target nodule(s) and near the planned trajectory of the biopsy instruments.
4. Presence of mediastinal nodal disease on pre-procedure CT or PET-CT scan.
5. Patient with American Society of Anesthesiologists Classification (ASA) ≥4.
6. Patient underwent a pneumonectomy.
7. Any invasive concomitant procedure (outside of lymph node staging) not related to the pulmonary nodule(s) or suspected disease state.
8. Female patient of child-bearing potential who is unable to take adequate contraceptive precautions or is known to be pregnant, and/or breast feeding.
9. Patient has a documented medical history of uncorrectable coagulopathy, bleeding, or platelet disorder.
10. Patient is taking antiplatelet or anticoagulant medications that cannot be stopped per standard practice.
11. Patient is currently participating or has participated in another Clinical Investigation within the past 30 days, such as interventional trials or trials with experimental agents or agents of unknown risk, that may affect the endpoints of this Clinical Investigation.
12. Investigator, in their professional opinion, has decided that it is in the patient's best interest to not participate in the Clinical Investigation.
13. Patient is not willing to comply with post study procedure participation requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield of sample(s) obtained (post learning curve) | Up to 13 months post procedure]
  Diagnostic yield is the number of nodules in which the procedure was diagnostic (either malignant or non-malignant), relative to the total number of attempted navigation procedures

SECONDARY OUTCOMES:
Sensitivity for malignancy of sample(s) obtained | Up to 13 months post procedure
  Sensitivity for malignancy of samples is assessed as the number of subjects with a malignant condition determined through the study procedure (true positives) relative to the number of subjects with an underlying malignant disease state (true positives + false negatives).
  The subjects underlying disease state will be determined by follow-up diagnostic interventions or treatment decisions/interventions, and/or radiographic follow-up.
Rate of achieving biopsy tool position within the targeted nodule(s) as confirmed by CBCT 3D imaging or the combination of multi-angle augmented fluoroscopy with diagnostic rapid onsite pathology (in the absence of a confirmatory spin). | At time of the biopsy procedure (Day 0)
  The rate of Tool in Nodule is how often the biopsy tool to sample the tissue is positioned directly within the nodule before the sample is taken.
  If biopsy forceps are used, it is how often the instrument is surrounding the nodule before the sample is taken.

OTHER OUTCOMES:
Rate of procedure-related Adverse Events through 7 days post-procedure | 7 days
  The study's safety endpoint is the rate of procedure-related Adverse Events through 7 days post-procedure
Procedure-related characteristics | At time of the biopsy procedure (Day 0)
  Procedure time (from catheter inserted into the patient's airways to catheter removed from the patient's airways) will be reported
rEBUS visualization characteristics | At time of the biopsy procedure (Day 0)
  The frequency of use of a concentric rEBUS visualization view during the biopsy will be summarized.
Biopsy workflow | At time of the biopsy procedure (Day 0)
  The sequence of biopsy tools used will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Sundeep Master, Study Director — Intuitive Surgical
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD.